CLINICAL TRIAL: NCT05781009
Title: Pregnenolone for the Treatment of Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000034929; R01AA030923 (NIH)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Pregnenolone

STUDY DESIGN:
Intervention Model Description: Randomized Double-blind, placebo-controlled, parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- patients receiving 300mg PREG (Active Comparator): Patients randomly assigned to receive 300mg of pregnenolone (PREG) daily.
  Interventions: Drug: Pregnenolone
- placebo (Placebo Comparator): Patients randomly assigned to receive a placebo daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — 300mg
  Arms: patients receiving 300mg PREG
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
This Phase 2 randomized cotrolled trial (RCT) will assess the safety and efficacy of pregnenolone (PREG; 300 mg/day, b.i.d dosing) vs. placebo (PBO) over a 12 week treatment period, and at 1-month post-treatment follow-up in individuals with Alcohol Use Disorder (AUD).

DETAILED DESCRIPTION:
In this Phase 2 single-site randomized controlled trial (RCT), men and women with Alcohol Use Disorder (AUD) will be enrolled in a 12 week trial with a 1-month follow-up assessment. Participants will be randomly assigned to 300mg pregnenolone (PREG) treatment b.i.d., or Placebo (PBO). All participants will be assessed 2x weekly and also receive behavior counseling to support recovery. The study aims to examine a) the safety and tolerability; b) efficacy on alcohol use outcomes; and c) effects on alcohol craving, anxiety, depression and physical well-being of 300mg PREG vs. PBO in men and women with AUD over the 12-week treatment period and at the 1-month follow up post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and females, aged 18-70 years;
* Regular weekly use of alcohol at least 3X weekly or more at treatment entry;
* Must meet current DSM-5 criteria for moderate to severe Alcohol Use Disorders (AUDs) using SCID-I for DSM-5;
* No health conditions that would impact trial participation as verified by screening and physical examination and absence of any of the exclusion criterions outlined below;
* Able to read English and complete study evaluations;
* Able to provide informed written and verbal consent.

Exclusion Criteria:

* Meet current criteria for moderate to severe substance use disorders from use of any other psychoactive substance, excluding nicotine and cannabis use disorder;
* Current use of opioids;
* Regular use of anticonvulsants, sedatives or hypnotics, oral prescription analgesics (other than non-steroidal anti-inflammatory drugs), topiramate, baclofen;
* Regular use of steroidal supplements and steroid medications interacting with study medications based on clinical judgement of study physician (excluding hormonal contraceptives in women);
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania);
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study, but stable, prescribed anti-hypertensives. cardiovascular and diabetes medications will be allowed after review by study physician;
* Any psychotic disorder or current Axis I psychiatric disorders requiring specific acute attention, including need for psychiatric medications, but stable, prescribed antidepressants and anti-anxiety medication to treat co-occurring psychiatric disorders will be allowed;
* Women who are pregnant, nursing or refuse to use a reliable form of birth control (as assessed by urine pregnancy tests during initial medical evaluation, and assessed every two weeks during the course of the study).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Percent of Subjects with no Heavy Drinking Days | 12 weeks
  Pregnenolone versus Placebo treated subjects will be compared on any days of heavy drinking which is defined by 5 or more drinks per day in men and 4 or more drinks/day in women. This will be measured by the Percent of Subjects with no Heavy Drinking Days (PSNHDD) over a 12 week period.
Safety of pregnenolone | 12 weeks
  The Systematic Assessment of Treatment Emergent Events (SAFTEE) Questionnaire will be used to assess adverse events weekly during the trial.

SECONDARY OUTCOMES:
Percent Heavy Drinking Days | 12 weeks
  Percent of overall days with heavy drinking days (defined by 5 or more drinks per day in men and 4 or more drinks/day in women).
Percent Any Drinking Days | 12 weeks
  Percent of any drinking days over a 12 week period.
Average Drinks per Day | 12 weeks
  The average number of drinks consumed per day assessed weekly over the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States